CLINICAL TRIAL: NCT01041274
Title: Citalopram in First Episode Schizophrenia
Brief Title: DECIFER: Depression and Citalopram In First Episode Recovery
Acronym: DECIFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-01965; 1R01MH084900-01A1 (NIH)
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia; Schizophreniform Disorder
Keywords: Schizophrenia; Citalopram; First episode; fMRI; Cognitive behavioral therapy; Psychoeducation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Citalopram; Dexetimide; Sugars; Therapeutics; Cognitive Behavioral Therapy; Neuroimaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram (Experimental): Participants will receive a daily dose of citalopram, with flexible dosing as determined by clinician, for 12 months.
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Participants will receive a daily dose of placebo for 12 months.
  Interventions: Drug: Placebo; Behavioral: Psychoeducation; Behavioral: Cognitive Behavioral Therapy (CBT); Radiation: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Drug: Citalopram — 40 mg by mouth daily for 12 months. Dosing will start at 20mg daily and may be increased after a minimum of one week to the target dose of 40 mg daily. Dose decreases will be made in the presence of side effects. Allowed dose range will be 10 mg daily to 40 mg daily.
  Other Names: Celexa; Cipramil
  Arms: Citalopram
Drug: Placebo — Placebo by mouth daily for 12 months.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Psychoeducation — 16 sessions of weekly, individual psychoeducation and relapse prevention planning followed by 8 monthly sessions
  Other Names: Therapy
  Arms: Placebo
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants who exhibit symptoms of moderate suicidality at any point during the trial will be treated with 12 sessions of CBT, either once or twice weekly based on clinical judgment. Participants who continue to exceed suicidality criteria after 4 weeks of CBT will be dropped from double-blind treatment and may be prescribed openly an SSRI
  Other Names: Therapy
  Arms: Placebo
Radiation: Functional Magnetic Resonance Imaging (fMRI) — 3 1-hour sessions of fMRI brain scanning, assessed at baseline, and weeks 24 and 52
  Other Names: Neuroimaging
  Arms: Placebo

SUMMARY:
This study seeks to examine the effectiveness of citalopram added to treatment with any oral or injectable second-generation antipsychotic plus standardized psychoeducation in first episode schizophrenia patients. Because depressive symptoms are common in first episode patients, we will test the hypothesis that adding the SSRI citalopram to a pre-established medication regimen will improve quality of life and decrease relapse and suicidality over the course of a 12-month trial.

DETAILED DESCRIPTION:
We propose to conduct a 12-month, placebo-controlled, double-blind, parallel-group trial of citalopram added to treatment with any oral or injectable second-generation antipsychotic plus standardized psychoeducation. Subjects will be 100 patients ages 16-40 with first episode schizophrenia or schizophreniform disorder with onset before age 35 who have received at least 4 weeks and fewer than 16 cumulative weeks of antipsychotic medication, have not been treated with an SSRI within four weeks and do not meet criteria for major depression or significant suicidal ideation. This study will be conducted by the Schizophrenia Program of the NYU Langone Medical Center and at the Psychiatry Outpatient Clinic of Bellevue Hospital located in New York, NY

Upon signing consent, patients will undergo screening procedures to assess eligibility. A diagnosis of schizophrenia or schizophreniform disorder will be determined by the Structured Clinical Interview for DSM IV (SCID) completed by a research clinician using all available clinical data and will be confirmed by consensus diagnosis. A comprehensive medical history and physical exam, including measurement of vital signs, will be performed. A psychiatric history, including diagnosis, treatment history, current medications, and substance use will also be performed. At screening only, a fasting blood sample will be obtained to perform routine laboratory tests including electrolytes, BUN, creatinine, liver function tests, fasting glucose, calcium, phosphate, magnesium, albumin and CBC with differential. Urinalysis will be performed to identify unstable medical illness. A urine toxicology screen will be performed and a urine pregnancy test will be done for women of child bearing potential. A research assistant will complete the demographics and administer the Calgary Depression Scale for Schizophrenia (CDSS), Scale for the Assessment of Negative Symptoms (SANS) and InterSePT Scale for Suicidal Thinking (ISST) to determine whether inclusion criteria are met.

Subjects who meet study eligibility criteria will complete the baseline assessment which will include the following assessments: Brief Psychiatric Rating Scale (BPRS), SANS, CDSS, ISST, Clinical Global Impression for Severity of Suicidality (CGI-SS), Clinical Global Impression (CGI), Heinrich Quality of Life Scale (QLS), WHO Quality of Life Scale (WHO-QOL), Scale for the Assessment of Positive Symptoms-Delusions (SAPS-D),Birchwood Insight Scale (IS), Brief Time Use Survey (BTUS), MIRECC Global Assessment of Functioning (MIRECC GAF), Beck Depression Inventory-II (BDI-II), State-Trait Anxiety Inventory (STAI),MacArthur Perceived Coercion Scale (PCS), Basis-24, Subject Well-being under Neuroleptic Scale (SWN-S),Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS), Brief Adherence Rating Scale (BARS), Medication Adherence Rating Scale (MARS), Social Behavior Scale (SBS), WHO Alcohol Smoking and Substance Involvement Screening Test (WHO ASSIST), and a Drug Use Survey. In addition, side effects will be rated using the Systematic Assessment for Treatment Emergent Events (SAFTEE), Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS) and the Simpson Angus Scale for Extrapyramidal Symptoms (SAS). Assessment of cognitive functioning will be measured by the MATRICS battery.

Subjects will undergo 4 high-resolution MP-RAGE scans: once each at Baseline, 2 months, 6 months and 12 months. Scheduled Participants will be randomized 1:1 to citalopram or placebo. We will follow a standard approach to flexible dosing with citalopram as recommended by the manufacturer, initiating treatment with a dose of 20 mg (two capsules) daily. Clinicians may increase or decrease the dose by one capsule every two weeks to a maximum of 4 capsules and a minimum of one capsule daily.

Beginning at Week 1, participants will receive 16 sessions of weekly, individual psychoeducation and relapse prevention planning followed by 8 monthly sessions. Participants who score 3 (moderate suicidality) on the CGI-SS or > 7 on the CDSS will be treated with a standard 12 session CBT approach to depression that includes elements targeting suicidality when appropriate. Clinical judgment will be used to determine whether to offer the CBT for depression sessions once or twice weekly.

The CDSS, ISST, and CGI-SS will be administered at baseline and then weekly up to week 8, then monthly. The SANS, BPRS, and BARS will be administered at baseline, then monthly for the duration of the study. The Heinrich's QOL and WHO QOL will be administered at baseline, and then monthly until study completion, excepting week 28, week 36, week 44, and week 48. The SAPS-D,IS, BTUS, MIRECC GAF, CGI, STAI, PCS, Basis-24, SWN-S, SSTICS, MARS, and SBS will be administered at baseline, week 24, and week 52. The BDI-II will be administered at screening, baseline, weeks 1-16, then monthly. The WHO-ASSIST will be administered at baseline, week 12, week 24, and week 52. The drug use survey will be administered at baseline, week 4, week 8, week 12, week 16, week 20, week 24, and week 52.

A fasting blood sample will be drawn at Baseline, weeks 4 and 8 and every 8 weeks thereafter for BDNF assay. Blood samples collected at Baseline, week 24, and week 52 will be assayed for prolactin and inflammation markers. Blood samples collected at baseline, week 8, week 24, and week 52 will be assayed for C-Reactive Protein. Additionally, a blood sample for DNA will be collected at week 4. Saliva will be collected with tongue swabs at Baseline, Week 4, Week 8, Week 16, Week 24, Week 36, and Week 52 for cortisol analyses.

Participants who choose to discontinue study drug will be asked if they are willing to continue their scheduled assessments. These subjects will continue to be followed for the entire course of the study but will not receive any study medication. Final study visit will be conducted 1 year post randomization.

The primary outcome measure is change in depression symptoms as measured by the Calgary Depression Scale total score. Secondary outcome measures include a measure of changes in negative symptoms (SANS), relapse rates (BPRS), suicidal ideation (ISST), and quality of life (QOL), measured at various time points during the 12-month trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 16-40 years
* Schizophrenia, any subtype or Schizophreniform disorder
* Treated with any of the following second generation antipsychotics for at least 4 weeks and fewer than 16 weeks: risperidone, olanzapine, quetiapine, aripiprazole, ziprasidone, or paliperidone)
* Willing to participate in psychoeducation
* Sufficient proficiency in English to complete assessments

Exclusion Criteria:

* Major depression by DSM-IV criteria
* Clinical Global Assessment of Severity of Suicidality of 3 (moderate) or greater.
* Calgary Depression Scale for Schizophrenia (CDRS) score of 7 or greater
* Serious suicide attempt within three years or ANY suicide attempt for subjects age 16-25.
* Current treatment with an MAOI or pimozide
* Active alcohol or other substance abuse or dependence within three months
* Unstable medical illness
* History of SSRI intolerance
* Pregnant or nursing
* QTc ≥ 500 msec

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center/ Bellevue Hospital, New York, New York, United States

REFERENCES:
- [Derived] Wang J, Hart KL, Qi W, Ardekani BA, Li C, Marx J, Freudenreich O, Cather C, Holt D, Bello I, Diminich ED, Tang Y, Worthington M, Zeng B, Wu R, Fan X, Zhao J, Wang J, Goff DC. Association of Aripiprazole With Reduced Hippocampal Atrophy During Maintenance Treatment of First-Episode Schizophrenia. J Clin Psychopharmacol. 2021 May-Jun 01;41(3):244-249. doi: 10.1097/JCP.0000000000001391. PMID 33814546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Citalopram | Placebo
Started (Total Randomized) | 49 | 46
Completed (Week 52 Completers) | 26 | 25
Not Completed | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram | Placebo | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.2 (5.09) | 23.69 (4.63) | 23.44 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 32 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 23 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Calgary Depression Scale for Schizophrenia (CDSS)
Description: The Calgary Depression Scale for Schizophrenia (CDSS) is a rater-administered assessment that measures depression in schizophrenia. The scale consists of 9 questions each rated 0 to 3. 0 corresponds with "absent" and 3 corresponds with "severe". The total score for all items is provided for each time point. The minimum score is 0 and the maximum score is 27. A higher score indicates increased depressive symptoms.
Time Frame: Screening, Baseline, Weeks 1-8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Not all participants completed the CDRS assessment at each time point. Results are reported for all participants who completed the CDRS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 49 | 46
units on a scale
  Screening: number analyzed (Participants) | 46 | 43
  Screening | 1.93 (1.74) | 2.26 (1.74)
  Baseline: number analyzed (Participants) | 46 | 45
  Baseline | 1.83 (1.79) | 2.58 (2.99)
  Week 1: number analyzed (Participants) | 16 | 17
  Week 1 | 2.13 (2.47) | 1.94 (3.03)
  Week 2: number analyzed (Participants) | 38 | 32
  Week 2 | 2.00 (2.34) | 1.84 (2.53)
  Week 3: number analyzed (Participants) | 20 | 15
  Week 3 | 2.4 (2.80) | 1.87 (2.53)
  Week 4: number analyzed (Participants) | 44 | 38
  Week 4 | 1.34 (1.95) | 1.79 (1.79)
  Week 5: number analyzed (Participants) | 13 | 12
  Week 5 | 1.54 (2.11) | 1.67 (1.78)
  Week 6: number analyzed (Participants) | 14 | 15
  Week 6 | 1.29 (1.54) | 1.07 (1.34)
  Week 7: number analyzed (Participants) | 15 | 13
  Week 7 | 1.20 (1.32) | 2.15 (2.76)
  Week 8: number analyzed (Participants) | 40 | 37
  Week 8 | 1.08 (2.27) | 1.49 (1.82)
  Week 12: number analyzed (Participants) | 39 | 34
  Week 12 | 1.41 (2.48) | 1.32 (2.03)
  Week 16: number analyzed (Participants) | 36 | 32
  Week 16 | .97 (1.44) | .72 (1.22)
  Week 20: number analyzed (Participants) | 35 | 31
  Week 20 | 1.11 (2.06) | 1.23 (1.61)
  Week 24: number analyzed (Participants) | 37 | 35
  Week 24 | 1.32 (1.89) | 1.20 (1.61)
  Week 28: number analyzed (Participants) | 30 | 29
  Week 28 | .67 (1.27) | 1.14 (1.30)
  Week 32: number analyzed (Participants) | 28 | 27
  Week 32 | .71 (1.12) | .81 (1.33)
  Week 36: number analyzed (Participants) | 26 | 31
  Week 36 | .42 (.86) | 1.06 (1.29)
  Week 40: number analyzed (Participants) | 26 | 29
  Week 40 | .96 (1.69) | 1.21 (1.93)
  Week 44: number analyzed (Participants) | 24 | 29
  Week 44 | .63 (1.53) | 1.55 (1.76)
  Week 48: number analyzed (Participants) | 24 | 23
  Week 48 | .5 (.89) | 1.3 (1.72)
  Week 52: number analyzed (Participants) | 25 | 27
  Week 52 | .4 (1.08) | 1.15 (1.68)

2. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: The Scale for the Assessment of Negative Symptoms (SANS) is a 25-item rater-administered scale to assess negative symptoms in schizophrenia. Each item is rated from 0 to 5 where 0 is "none" and 5 is "severe". The SANS consists of five subscales: affective flattening/blunting, alogia, avolition/apathy, ahnedonia/asociality, and attention. Each subscale contains a "global rating" item which assesses the overall severity of symptoms within the subscale. The total score consists of a sum of all items except the global ratings and items 10, 23, 24, and 25. The total score is reported for each time point. The minimum total score is 0 and the maximum total score is 85. A higher score indicates increased severity of negative symptoms.
Time Frame: Screening, Baseline, Weeks 4, 8, 12, 16, 20, 24, 28,32, 36, 40, 44, 48, 52
Population: Not all participants completed the SANS assessment at each time point. Results are reported for all participants who completed the SANS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 49 | 46
units on a scale
  Screening: number analyzed (Participants) | 46 | 43
  Screening | 19.89 (14.39) | 16.77 (11.9)
  Baseline: number analyzed (Participants) | 46 | 45
  Baseline | 21.37 (14.25) | 18.91 (12.08)
  Week 4: number analyzed (Participants) | 44 | 38
  Week 4 | 16.98 (14.17) | 14.58 (10.23)
  Week 8: number analyzed (Participants) | 40 | 37
  Week 8 | 13.83 (12.04) | 13.11 (10.58)
  Week 12: number analyzed (Participants) | 39 | 34
  Week 12 | 12.38 (12.21) | 14.06 (11.73)
  Week 16: number analyzed (Participants) | 36 | 33
  Week 16 | 11.08 (11.34) | 11.48 (10.14)
  Week 20: number analyzed (Participants) | 34 | 31
  Week 20 | 12.26 (13.10) | 12.29 (11.78)
  Week 24: number analyzed (Participants) | 37 | 36
  Week 24 | 12.41 (12.06) | 13.06 (11.23)
  Week 28: number analyzed (Participants) | 29 | 29
  Week 28 | 9.9 (11.04) | 12.59 (11.71)
  Week 32: number analyzed (Participants) | 28 | 26
  Week 32 | 8.0 (9.15) | 10.92 (10.77)
  Week 36: number analyzed (Participants) | 26 | 31
  Week 36 | 8.38 (9.76) | 11.68 (10.62)
  Week 40: number analyzed (Participants) | 26 | 28
  Week 40 | 9.35 (11.93) | 10.64 (12.67)
  Week 44: number analyzed (Participants) | 24 | 28
  Week 44 | 7.54 (8.92) | 12.64 (12.98)
  Week 48: number analyzed (Participants) | 24 | 23
  Week 48 | 7.54 (9.10) | 13.0 (13.88)
  Week 52: number analyzed (Participants) | 26 | 25
  Week 52 | 13.83 (12.04) | 11.64 (13.92)

3. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The Brief Psychiatric Rating Scale (BPRS) is a 24-item rater-administered scale assessing overall psychiatric and psychotic symptoms. Items 1-14 are assessed through self-report and items 15-24 are assessed on the basis of observed behavior. Each item is rated from 1 to 7 where 1 is "not present" and 7 is "extremely severe". A score of 0 indicates "not assessed". The total score is a sum of all items and is reported for each time point. The minimum score is 24 and the maximum score is 168, and higher values indicate increased symptom severity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Not all participants completed the BPRS assessment at each time point. Results are reported for all participants who completed the BPRS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 49 | 46
units on a scale
  Baseline: number analyzed (Participants) | 46 | 45
  Baseline | 39 (11.5) | 38.0 (9.3)
  Week 4: number analyzed (Participants) | 44 | 38
  Week 4 | 33.11 (7.3) | 33.1 (6.7)
  Week 8: number analyzed (Participants) | 40 | 37
  Week 8 | 33.3 (9.2) | 33.2 (8.0)
  Week 12: number analyzed (Participants) | 40 | 34
  Week 12 | 33.8 (10.0) | 33.2 (7.2)
  Week 16: number analyzed (Participants) | 22 | 19
  Week 16 | 27.9 (5.9) | 29.1 (4.9)
  Week 20: number analyzed (Participants) | 35 | 31
  Week 20 | 33.1 (9.9) | 31.2 (7.5)
  Week 24: number analyzed (Participants) | 38 | 35
  Week 24 | 32.6 (9.8) | 32.7 (7.6)
  Week 28: number analyzed (Participants) | 30 | 29
  Week 28 | 29.6 (5.5) | 31.6 (7.3)
  Week 32: number analyzed (Participants) | 28 | 27
  Week 32 | 29.4 (5.5) | 29.9 (5.6)
  Week 36: number analyzed (Participants) | 26 | 31
  Week 36 | 28.6 (5.3) | 32.2 (9.7)
  Week 40: number analyzed (Participants) | 26 | 28
  Week 40 | 31.1 (7.7) | 31.4 (8.3)
  Week 44: number analyzed (Participants) | 24 | 28
  Week 44 | 30.1 (7.9) | 33.5 (10.1)
  Week 48: number analyzed (Participants) | 24 | 23
  Week 48 | 30.0 (6.7) | 32.6 (9.0)
  Week 52: number analyzed (Participants) | 26 | 26
  Week 52 | 29.1 (6.9) | 32.7 (11.2)

4. Secondary Outcome: InterSePT Scale for Suicidal Thinking (ISST)
Description: IntraSePT Scale for Suicidal Thinking (ISST) consists of 12 questions rated from 0 to 2 with increasing intensity (i.e. none, weak, moderate to stron). It quantifies the current conscious and overtly expressed suicidal thinking in schizophrenic patients by canvassing various suicidal thoughts and wishes during a 20- to 30-min semi-structured interview. The total score is computed by adding the 12 individual item scores and ranges from 0 to 24. A score of zero indicates low suicidal ideation and a score of 24 indicates high suicidal ideation.
Time Frame: Screening, Baseline, Weeks 1-8
Population: Given the low scores on this assessment, data collection was discontinued.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 49 | 46
score on a scale
  Screening: number analyzed (Participants) | 25 | 24
  Screening | 0.184 (0.808) | 0.643 (2.57)
  Baseline: number analyzed (Participants) | 43 | 39
  Baseline | 0.605 (1.76) | 0.462 (1.57)
  Week 1: number analyzed (Participants) | 18 | 19
  Week 1 | 0.667 (2.14) | 0.263 (0.806)
  Week 2: number analyzed (Participants) | 41 | 24
  Week 2 | 0.293 (1.585) | 0.0 (0.0)
  Week 3: number analyzed (Participants) | 22 | 16
  Week 3 | 0.136 (0.640) | 1.00 (3.29)
  Week 4: number analyzed (Participants) | 47 | 27
  Week 4 | 0.0 (0.0) | 0.0 (0.0)
  Week 5: number analyzed (Participants) | 14 | 13
  Week 5 | 0.357 (1.34) | 0.0 (0.0)
  Week 6: number analyzed (Participants) | 16 | 16
  Week 6 | 0.125 (0.50) | 0.0 (0.0)
  Week 7: number analyzed (Participants) | 18 | 14
  Week 7 | 0.0 (0.0) | 0.0 (0.0)
  Week 8: number analyzed (Participants) | 42 | 25
  Week 8 | 0.0 (0.0) | 0.20 (0.816)

5. Secondary Outcome: Heinrich Quality of Life Scale (QOL)
Description: The Quality of Life Scale (QOL) is a 21-item scale based on a semi-structured interview to assess functional deficits in schizophrenia. Each item is rated on a 7-point scale where 0 indicates a normal level of functioning, or no deficit, and 6 corresponds to more severe deficit. The total score is a sum of all items. The minimum total score is 0 and the maximum total score is 126, higher scores indicate increased impairment in functioning.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 32, 40, 52
Population: Not all participants completed the QOL assessment at each time point. Results are reported for all participants who completed the QOL assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 49 | 46
units on a scale
  Baseline | 71.5 (25.9) | 75.9 (23.2)
  Week 4: number analyzed (Participants) | 47 | 39
  Week 4 | 81.0 (24.3) | 83.6 (21.8)
  Week 8: number analyzed (Participants) | 42 | 38
  Week 8 | 86.2 (25.2) | 87.1 (21.1)
  Week 12: number analyzed (Participants) | 41 | 35
  Week 12 | 86.4 (27.9) | 90.4 (22.7)
  Week 16: number analyzed (Participants) | 38 | 34
  Week 16 | 89.6 (27.8) | 92.1 (20.0)
  Week 20: number analyzed (Participants) | 37 | 32
  Week 20 | 86.4 (29.6) | 91.8 (23.4)
  Week 24: number analyzed (Participants) | 39 | 37
  Week 24 | 87.4 (28.8) | 92.9 (20.3)
  Week 32: number analyzed (Participants) | 28 | 28
  Week 32 | 98.7 (26.0) | 98.0 (21.4)
  Week 40: number analyzed (Participants) | 26 | 30
  Week 40 | 100.2 (25.3) | 91.1 (29.6)
  Week 52: number analyzed (Participants) | 26 | 27
  Week 52 | 86.2 (25.2) | 95.6 (28.6)

ADVERSE EVENTS:
Description: Non-serious adverse events were reported through the Systematic Assessment of Treatment Emergent Effects (SAFTEE) questionnaire unless otherwise specified.
Arm/Group | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 5/49 | 4/46
Other Adverse Events (participants affected / at risk) | 22/49 | 18/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=49) | Placebo (N=46)
Psychiatric Hospitalization (Psychiatric disorders) | 3 (4) | 4 (4) — Hospitalization for worsening symptoms of psychosis including paranoia, suicidal ideation, homicidal ideation, and/or auditory and visual hallucinations.
Incarceration (Psychiatric disorders) | 1 (1) | 1 (1) — Patient incarcerated during study
Medical Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Pneumonia
Drug-related hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=49) | Placebo (N=46)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorgasmia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 2 (2)
Appetite decrease (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Appetite increase (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Concentration impaired (Psychiatric disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Emotional dejection (Psychiatric disorders) | 0 (0) | 1 (1)
Difficulty thinking (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness upon standing (Nervous system disorders) | 1 (1) | 1 (4)
Drooling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (2) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 2 (2)
Faintness (Nervous system disorders) | 0 (0) | 1 (1)
False sensation (Nervous system disorders) | 0 (0) | 2 (2)
Fatigue (Nervous system disorders) | 1 (3) | 2 (2)
Hiccup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hit by a motorcycle (General disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hurt when riding a bike (General disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Loss of libido (Reproductive system and breast disorders) | 3 (6) | 1 (1)
Memory impaired (Nervous system disorders) | 2 (2) | 1 (4)
Mental activity decreased (Nervous system disorders) | 1 (1) | 1 (1)
Muscle twitch (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Restlessness (Nervous system disorders) | 2 (2) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 2 (8) | 1 (2)
Sleeplessness (Nervous system disorders) | 1 (1) | 1 (1)
Taste alteration (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Weight increase (Metabolism and nutrition disorders) | 9 (9) | 6 (7)
Sensory hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disturbed (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Vascular disorders) | 5 (10) | 0 (0)
Teeth grating (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No